CLINICAL TRIAL: NCT07277205
Title: Comparison of the Effects of Vestibular Rehabilitation and Dual-Task Exercise Programs on Cognitive and Motor Functions in Individuals With Parkinson's Disease
Brief Title: Comparison of Vestibular and Dual-Task Rehabilitation in Parkinson's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ezgi Eryıldız, Research assistant, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09.2025.304
Record Dates: First submitted 2025-11-20; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vestibular Rehabilitation Group (Experimental)
  Interventions: Other: Vestibular Rehabilitation
- Cognitive-Motor Dual Task Activities Group (Experimental)
  Interventions: Other: Cognitive-Motor Dual Task Activities
- Control Group (No Intervention)

INTERVENTIONS:
Other: Vestibular Rehabilitation — Vestibular exercises will consist of static and dynamic balance exercises, VOR and eye movement training, central balance strategies and static-dynamic balance, adaptation, substitution, habituation exercises in terms of adapting to the balance system.
  Arms: Vestibular Rehabilitation Group
Other: Cognitive-Motor Dual Task Activities — In the Cognitive-Motor Dual Task Activities Group, patients will be given additional cognitive tasks (e.g. counting months, subtracting 5 from 100, etc.) in line with the physiotherapist's commands simultaneously with balance and functional activities (such as stepping forwards-sideways-backwards, sitting-standing).
  Arms: Cognitive-Motor Dual Task Activities Group

SUMMARY:
Parkinson's disease (PD) is a long-term condition that affects movement, balance, and thinking abilities. It can cause tremor, stiffness, slow movements, and difficulty maintaining balance. In addition to these physical problems, many people with PD also experience difficulties with memory, attention, and other cognitive functions. The balance system in the inner ear (vestibular system) helps maintain posture and orientation, but this system may not work properly in people with PD.

This study aims to compare two different types of exercise programs to improve movement, balance, and cognitive abilities in individuals with PD. One program focuses on exercises that stimulate the balance system (vestibular rehabilitation), while the other combines thinking and movement activities at the same time (dual-task training).

Thirty-six people with PD will take part in the study. Participants will be randomly assigned to one of three groups: vestibular exercise group, dual-task exercise group, or control group. Exercises will be done under the supervision of a physiotherapist twice a week for eight weeks. Each session will last about 40 minutes and include activities that are safe, structured, and personalized.

Before and after the 8-week program, participants will complete simple tests that measure their memory, attention, walking ability, balance, and daily activity level. The results will show whether these exercise approaches can help improve both body and brain functions.

The findings of this study are expected to help physiotherapists design more effective and personalized rehabilitation programs for people with Parkinson's disease, leading to better balance, safer movement, and improved quality of life.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a chronic, progressive neurodegenerative disorder characterized by motor symptoms such as tremor, rigidity, bradykinesia, and postural instability, as well as non-motor symptoms including cognitive impairment and depression. Postural control depends on the integration of visual, somatosensory, and vestibular inputs, and this multisensory integration is often impaired in PD. Vestibular dysfunction can manifest as dizziness, imbalance, and spatial disorientation, leading to functional limitations, an increased risk of falls, and reduced independence. Moreover, the vestibular system is anatomically and functionally connected to brain regions involved in cognition, such as the hippocampus and frontal cortex. Therefore, targeting vestibular function in rehabilitation may improve not only balance but also cognitive performance.

Previous research has demonstrated that vestibular rehabilitation can improve balance, gait, and postural stability in individuals with PD. However, its potential effects on cognitive functions have been largely neglected. In parallel, dual-task training-based on the simultaneous performance of motor and cognitive tasks-has emerged as an evidence-based approach to improve both motor and cognitive outcomes. Studies have shown that dual-task exercise can enhance gait speed, step length, balance, attention, and executive function in PD. Nevertheless, no studies have directly compared the effects of vestibular rehabilitation and dual-task exercise training on cognitive and motor functions in this population.

The present study is designed to fill this gap by comparing these two rehabilitation approaches. A total of 36 participants diagnosed with PD will be recruited and randomly assigned into three groups: (1) vestibular rehabilitation, (2) cognitive-motor dual-task training, and (3) control. Each intervention will be administered twice weekly for eight weeks, with each session lasting approximately 40 minutes under the supervision of a physiotherapist. The vestibular rehabilitation program will include static and dynamic balance training, gaze stabilization, adaptation, habituation, and substitution exercises. The dual-task training program will integrate functional balance exercises with concurrent cognitive challenges (e.g., counting backward, naming tasks, or alternating verbal tasks). The control group will maintain their usual level of physical activity.

Assessments will be conducted before and after the 8-week intervention. Cognitive functions will be evaluated using the Digit Span Test, Word Fluency Test, and Clock Drawing Test. Motor functions will be assessed with the Mini-BESTest, Four Square Step Test, and Dynamic Gait Index, along with postural stability analysis using KFORCE Plates. Activity and participation will be evaluated using the Parkinson's Activity Scale and the Parkinson's Disease Questionnaire (PDQ-39).

Data will be analyzed using SPSS 21.0. Depending on normality assumptions, repeated-measures ANOVA or non-parametric alternatives will be used to assess within- and between-group differences. Statistical significance will be set at p < 0.05.

This study is expected to provide new insights into the clinical impact of vestibular and dual-task rehabilitation on cognitive and motor outcomes in PD. The results may contribute to developing individualized, evidence-based physiotherapy protocols that integrate balance and cognitive training, ultimately improving functional independence and quality of life among individuals with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 40 and 75 years
* Diagnosed with idiopathic Parkinson's disease (IPD)
* Stable medication regimen within the past one month
* Hoehn and Yahr stage I-III
* A score of at least 22 on the Montreal Cognitive Assessment (MoCA)
* Participants evaluated during the "on" phase of their medication cycle
* No hearing and/or visual impairments

Exclusion Criteria:

* Presence of any neurological, cardiovascular, or orthopedic disorder that may interfere with walking
* Diagnosis of any other neurological disease (e.g., dementia, cerebrovascular disease)
* Patients with deep brain stimulation (DBS) implants
* Presence of vascular pathologies in the lower extremities

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Mini-BESTest Total Score | Baseline and Week 8
  Dynamic balance will be assessed using the Mini-BESTest, consisting of 14 items scored from 0-2. The total score (0-28) will be used as the primary outcome, with higher scores indicating better balance and postural control.
  Unit of Measure: Points (0-28)
Semantic Verbal Fluency Test (Semantic Fluency, 60 seconds) | Baseline and Week 8
  Participants will name as many semantic-category words as possible within 60 seconds. The outcome will be the total number of correct words produced.
  Unit of Measure: Number of words

SECONDARY OUTCOMES:
Digit Span Test (Forward and Backward) | Baseline and Week 8
  Attention and working memory will be evaluated using the Digit Span Test. Numbers are read at one-per-second pace, and participants repeat increasingly longer sequences forward and backward. Outcome: maximum correctly recalled span for each condition.
  Unit of Measure: Digit span (number of digits)
Clock Drawing Test (Manos & Wu Scoring Method) | Baseline and Week 8
  Visuospatial and executive functions will be assessed by drawing "10 past 11" on a pre-segmented circle. Correct placement of 8 numbers and 2 clock hands are scored. Total score ranges from 0 to 10.
  Unit of Measure: Points (0-10)
Four Square Step Test (FSST) | Baseline and Week 8
  Participants step clockwise and counterclockwise through four squares following a fixed sequence. Time to complete the sequence is recorded. The best of two trials will be used.
  Unit of Measure: Seconds
Dynamic Gait Index (DGI) Total Score | Baseline and Week 8
  Dynamic balance during gait will be assessed using the Dynamic Gait Index. Eight items are scored from 0-3, with a maximum score of 24. Higher scores indicate better performance.
  Unit of Measure: Points (0-24)
Postural Stability (KFORCE Plates - Center of Pressure Metrics) | Baseline and Week 8
  Static and dynamic balance parameters (e.g., center-of-pressure displacement, sway, weight distribution) will be recorded using KFORCE force plates. Objective biomechanical data will be extracted from standardized stance and movement conditions.
  Unit of Measure: Center of pressure metrics (mm or mm/s)
Parkinson Activity Scale (PAS) Total Score | Baseline and Week 8
  Functional mobility and activity performance will be assessed using the Parkinson Activity Scale. Scores range from 0 to 4 for each item, with higher scores indicating better functional ability.
  Unit of Measure: Points
Parkinson's Disease Quality of Life Questionnaire (PDQ-39) Total Score | Baseline and Week 8
  Quality of life will be measured with the PDQ-39, a 39-item questionnaire evaluating mobility, daily activities, emotional well-being, cognition, communication, and social functioning. Scores range 0-100, with higher scores indicating poorer quality of life.
  Unit of Measure: Total score (0-100)

IPD SHARING:
Plan to Share IPD: No